CLINICAL TRIAL: NCT04227964
Title: Periodontal Regeneration vs Extraction and Replacement of Teeth Severely Compromised by Attachment Loss to the Apex: a 10-year RCT
Brief Title: Periodontal Regeneration Versus Tooth Extraction and Replacement Denture in Teeth With Periodontal Hopeless Prognosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The European Research Group on Periodontology (ERGOPerio) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATRO1998
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Periodontitis Complex
Keywords: periodontitis; periodontal regeneration; tooth extraction; dental implant; fixed partial denture; survival analysis; Complication free survival; Recurrence analysis; Oral health related quality of life
MeSH Terms: conditions — Periodontitis | interventions — Tooth Extraction; Replantation

STUDY DESIGN:
Intervention Model Description: Single center RCT
Who Masked: Outcomes Assessor
Masking Description: Independent examiner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontal regeneration (Experimental): Periodontal regeneration consisting of papilla preservation flaps, application of FDA approved CE marked periodontal regenerative devices, tooth splinting and root canal treatment as required.
  Interventions: Device: Enamel matrix derivative, bone replacement graft, barrier membrane
- Extraction and tooth replacement (Active Comparator): Tooth extraction and replacement with a dental implant or a fixed partial denture following healing and reconstruction of the extraction area. Choice based on standard of practice.
  Interventions: Procedure: Tooth extraction and replacement

INTERVENTIONS:
Device: Enamel matrix derivative, bone replacement graft, barrier membrane
  Arms: Periodontal regeneration
Procedure: Tooth extraction and replacement
  Arms: Extraction and tooth replacement

SUMMARY:
Periodontal regeneration can change tooth prognosis and represents an alternative to extraction in teeth compromised by severe intrabony defects. The aim of this study is to compare periodontal regeneration (PR) with tooth extraction and replacement (TER) in a population with attachment loss to or beyond the apex of the root in terms of professional, patient reported and economic outcomes.

DETAILED DESCRIPTION:
This was a single center 10-year randomized controlled clinical trial. 50 stage III or IV periodontitis subjects with a severely compromised tooth with attachment loss to or beyond the apex were randomized to PR or TER with either an implant or a tooth supported fixed partial denture. Subjects were kept on a strict periodontal supportive care regimen every 3 months and examined yearly. Survival, complication free survival, recurrence analysis, oral health related quality of life and patient reported outcomes analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Non-smokers or smokers with less than 20/day
* Good oral hygiene (FMPS<25%)
* Good control of periodontitis (FMBS<25%)
* Good compliance with treatment
* Presence of generalised stage III or IV periodontitis
* Radiographic bone loss to the apex or beyond the apex of the root at at least one interdental aspect
* Presence of severe clinical attachment level loss (>10 mm)
* Presence of clearly identifiable crest of bone in adjacent teeth
* Lack of function due to hyper mobility
* Vital or non-vital teeth

Exclusion Criteria:

* Medical contraindication to elective surgery
* Poor oral hygiene
* Incomplete control of periodontitis in the dentition
* Inadequate compliance
* Inability to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 1998-06-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Tooth or tooth replacement survival | 10 year
  Presence of functional and symptoms free tooth or tooth replacement
Occurrence and cost of management of recurrence | 10-year
  Recurrence analysis
Oral health related quality of life: OHIP-14 (Oral Health Impact Profile) | 10 years
  14 validated questions, 5 point Liker scale, smaller scores represent better outcome (smaller impact on quality of life)

SECONDARY OUTCOMES:
Clinical attachment level gain | 10 years
  Control outcome of periodontal regeneration
Probing pocket depth | 10 years
  Control outcome of periodontal regeneration

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Cortellini, MD, Study Director — Investigator
Locations (1):
- Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cortellini P, Stalpers G, Mollo A, Tonetti MS. Periodontal regeneration versus extraction and dental implant or prosthetic replacement of teeth severely compromised by attachment loss to the apex: A randomized controlled clinical trial reporting 10-year outcomes, survival analysis and mean cumulative cost of recurrence. J Clin Periodontol. 2020 Jun;47(6):768-776. doi: 10.1111/jcpe.13289. Epub 2020 Apr 19. PMID 32249446